CLINICAL TRIAL: NCT07276906
Title: A Prospective, Randomized, Double-Blind, Non-Inferiority Trial Comparing Intramuscular Fentanyl and Ketorolac With Nerve of Arnold Block for Postoperative Pain Management in Pediatric Patients Undergoing Bilateral Myringotomy With Tympanostomy Tube Placement
Brief Title: Comparing Intramuscular Fentanyl and Ketorolac With Nerve of Arnold (NOA) Block for Bilateral Myringotomy
Acronym: NOA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of South Alabama (Other)
Responsible Party: Principal Investigator, Karthik Swamy, Director, Pediatric Anesthesiology, Principal Investigator, Assistant Professor, University of South Alabama
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2387143-1
Record Dates: First submitted 2025-11-19; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Fentanyl; Ketorolac; Ketorolac Tromethamine; Dexmedetomidine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IM Arm standard Care (Active Comparator): Patients receive intramuscular fentanyl 2 mcg/kg (maximum 100 mcg) plus intramuscular ketorolac 0.5 mg/kg (maximum 30 mg) after induction of anesthesia. Sham bilateral Nerve of Arnold block with normal saline 0.2 mL per side is performed to maintain blinding.
  Interventions: Drug: Fentanyl; Drug: Ketorolac; Procedure: Sham Nerve of Arnold Block
- Nerve block arm (Experimental): Patients receive bilateral Nerve of Arnold block with bupivacaine 0.25% with epinephrine 1:200,000 (0.2 mL per side) plus dexmedetomidine 5 mcg per side (maximum total bupivacaine dose 2.5 mg/kg) after induction of anesthesia. sham intramuscular injection with normal saline is performed to maintain blinding.
  Interventions: Procedure: Nerve of Arnold Block; Procedure: Sham Intramuscular Injection; Drug: Dexmedetomidine; Drug: Bupivacaine

INTERVENTIONS:
Drug: Fentanyl — Intramuscular fentanyl 2 mcg/kg (maximum 100 mcg) administered after induction of anesthesia
  Arms: IM Arm standard Care
Drug: Ketorolac — Intramuscular ketorolac 0.5 mg/kg (maximum 30 mg) administered after induction of anesthesia
  Other Names: Toradol
  Arms: IM Arm standard Care
Procedure: Nerve of Arnold Block — Bilateral Nerve of Arnold block with bupivacaine 0.25%, 0.2 mL per side (total 0.4 mL), administered after induction of anesthesia
  Arms: Nerve block arm
Procedure: Sham Intramuscular Injection — sham intramuscular injections with normal saline to maintain blinding
  Arms: Nerve block arm
Procedure: Sham Nerve of Arnold Block — Bilateral sham Nerve of Arnold block with normal saline 0.2 mL per side to maintain blinding
  Arms: IM Arm standard Care
Drug: Dexmedetomidine — Dexmedetomidine 5 mcg per side (10 mcg total) added to bupivacaine solution for Nerve of Arnold block as adjuvant to prolong block duration
  Other Names: Precedex
  Arms: Nerve block arm
Drug: Bupivacaine — Bupivacaine 0.25% with epinephrine 1:200,000, 0.2 mL per side (total 0.4 mL, maximum 2.5 mg/kg) for bilateral Nerve of Arnold block
  Other Names: Marcaine, Sensorcaine
  Arms: Nerve block arm

SUMMARY:
Background: Bilateral myringotomy with tympanostomy tube (BMT) placement is one of the most common pediatric surgical procedures. Despite its brief duration, many children experience significant postoperative pain. Current standard care typically involves intramuscular (IM) administration of an opioid (fentanyl) combined with a non-steroidal anti-inflammatory drug (ketorolac). While this multimodal approach provides adequate pain control for approximately 75% of children, it is associated with opioid-related side effects including respiratory depression, nausea, vomiting, and sedation. Additionally, nearly one-quarter of children still experience moderate-to-severe pain despite this regimen.

The Nerve of Arnold block is a regional anesthesia technique that involves injection of local anesthetic near the auricular branch of the vagus nerve, which provides sensory innervation to the external auditory canal and tympanic membrane. This technique offers the potential for targeted, opioid-sparing analgesia with extended duration and minimal systemic side effects. However, high-quality evidence comparing this regional technique to standard systemic analgesia in pediatric patients is lacking.

Study Objective: This study aims to determine whether the Nerve of Arnold block is non-inferior to the standard combination of IM fentanyl and IM ketorolac in controlling postoperative pain in children undergoing BMT placement.

Study Design: This is a prospective, randomized, double-blind, non-inferiority trial. Three hundred children aged 6 months to 6 years scheduled for bilateral myringotomy with tympanostomy tube placement will be randomized 1:1 to receive either: (1) Standard care: IM fentanyl (1-2 mcg/kg) plus IM ketorolac (0.5 mg/kg) with sham Nerve of Arnold block, or (2) Intervention: Bilateral Nerve of Arnold block with bupivacaine 0.25% plus sham IM injections. Both patients and outcome assessors will be blinded to treatment assignments.

Primary Outcome: The proportion of patients experiencing moderate-to-severe pain (Face, Legs, Activity, Cry, Consolability [FLACC] scale score ≥4) in the Post-Anesthesia Care Unit (PACU). Non-inferiority will be declared if the upper bound of the 95% confidence interval for the difference in proportions is less than 10 percentage points.

Secondary Outcomes: Secondary outcomes include mean and maximum FLACC scores, rescue analgesic requirements, respiratory depression, postoperative nausea and vomiting, PACU length of stay, parent satisfaction, and pain at 24 hours postoperatively.

Clinical Significance: If the Nerve of Arnold block is shown to be non-inferior to standard care, it could provide a valuable opioid-sparing alternative for postoperative pain management in pediatric ear surgery, potentially reducing opioid-related adverse events while maintaining effective analgesia. This would be particularly beneficial for patients with contraindications to opioids or NSAIDs and aligns with national efforts to reduce opioid exposure in pediatric populations.

DETAILED DESCRIPTION:
Clinical Context Bilateral myringotomy with tympanostomy tube placement is performed in over 600,000 children annually in the United States for treatment of recurrent acute otitis media or chronic otitis media with effusion. Despite being a brief minimally invasive procedure, inadequate postoperative pain control is common and associated with emergence agitation, delayed discharge, increased rescue medication requirements, and parental anxiety.

Current Standard of Care Recent large retrospective cohort studies have established the efficacy of multimodal analgesia for pediatric myringotomy and tube placement. Combined intramuscular fentanyl and ketorolac resulted in approximately 23% of children experiencing moderate-to-severe pain in the Post-Anesthesia Care Unit, compared to over 50% with ketorolac alone. These findings support multimodal analgesia as the current standard but also highlight that nearly one in four children still experience inadequate pain control despite optimized systemic therapy.

Limitations of Current Approach The standard opioid-NSAID combination has several limitations: opioid-related side effects including respiratory depression, nausea, vomiting, and sedation; growing concerns about opioid exposure in children; NSAID contraindications in patients with renal impairment, bleeding disorders, or hypersensitivity; systemic distribution with potential for widespread effects; limited duration of action; and residual pain in high-risk subgroups such as younger children and those with normal middle ears.

Nerve of Arnold Block as Alternative The Nerve of Arnold, the auricular branch of the vagus nerve, provides sensory innervation to the posterior external auditory canal and tympanic membrane, which is the surgical site for myringotomy and tube placement. Blocking this nerve with local anesthetic offers theoretical advantages including opioid-sparing analgesia with elimination of opioid-related side effects, targeted analgesia directly at the surgical site, extended duration with long-acting local anesthetics, minimal systemic absorption and side effects, and applicability to patients with contraindications to systemic agents.

The technique involves subcutaneous injection of local anesthetic in the space between the mastoid process and the posterior wall of the external auditory canal. While anatomical studies support consistent nerve location and the block has been described in adult case reports, no randomized controlled trials have evaluated its efficacy and safety compared to standard care in pediatric patients.

Study Rationale There is a critical gap in high-quality evidence comparing regional anesthesia techniques to systemic analgesia for pediatric myringotomy and tube placement. This study addresses this gap and aligns with national priorities for opioid-sparing pain management strategies.

Study Design This is a prospective, randomized, double-blind, parallel-group, non-inferiority trial. Three hundred children aged 6 months to 6 years undergoing bilateral myringotomy with tympanostomy tube placement will be randomized in a 1:1 ratio to receive either standard care with intramuscular fentanyl and ketorolac or bilateral Nerve of Arnold block with bupivacaine. Randomization will use a computer-generated sequence with variable block sizes to prevent prediction of treatment assignment.

Blinding Strategy This is a double-blind study with patients, parents, anesthesiologists, surgeons, PACU nurses, and outcome assessors blinded to treatment assignment. Blinding is maintained through use of sham procedures. Patients in the standard care group receive sham Nerve of Arnold blocks with normal saline, while patients in the intervention group receive sham intramuscular injections with normal saline. Study medications are prepared and labeled by the investigational pharmacy with identical appearance.

Interventions Standard Care Group: Patients receive intramuscular fentanyl 2 micrograms per kilogram (maximum 100 micrograms) and intramuscular ketorolac 0.5 milligrams per kilogram (maximum 30 milligrams) administered after induction of anesthesia, plus sham bilateral Nerve of Arnold blocks with normal saline 0.2 milliliters per side.

Intervention Group: Patients receive bilateral Nerve of Arnold blocks with bupivacaine 0.25% solution with 1 in 200000 epinephrine ,0.2 milliliters per side with dexmedetomidine 5 mics per side as adjuvant, plus sham intramuscular injections with normal saline.

All patients receive standardized general anesthesia with sevoflurane and spontaneous ventilation via face mask or laryngeal mask airway. No additional intraoperative analgesics are administered beyond the study interventions.

Rescue Analgesia Protocol Rescue analgesia is available in the Post-Anesthesia Care Unit for patients with FLACC scale scores of 4 or greater, indicating moderate-to-severe pain. First-line rescue medication is oral acetaminophen 20 milligrams per kilogram. Second-line rescue is oral oxycodone 0.1 milligrams per kilogram or intravenous morphine 0.05 milligrams per kilogram for patients unable to take oral medications.

Non-Inferiority Margin The non-inferiority margin is set at 10 percentage points. This margin was selected based on clinical significance and risk-benefit considerations. An increase in the proportion with moderate-to-severe pain from approximately 23% to 33% would remain substantially better than historical controls with ketorolac alone and may be acceptable if offset by opioid-sparing benefits including reduced respiratory depression, nausea, vomiting, and sedation.

Sample Size A total of 300 patients will be enrolled, with 150 patients per group. This sample size provides 80% power to detect non-inferiority with a one-sided alpha of 0.025, assuming a baseline rate of 23.5% in the standard care group, an anticipated rate of 25-28% in the intervention group, and accounting for 10% dropout or protocol violations.

Statistical Analysis The primary analysis will use an intention-to-treat approach comparing the proportion of patients with FLACC scores of 4 or greater between groups. Non-inferiority will be declared if the upper bound of the one-sided 97.5% confidence interval for the difference in proportions (intervention minus standard care) is less than 10 percentage points. A per-protocol analysis will be conducted as a sensitivity analysis. Secondary outcomes will be analyzed using appropriate statistical tests including t-tests, chi-square tests, and multivariable regression models. Subgroup analyses will explore effect modification by age group and middle ear condition.

Safety Monitoring All patients will have continuous monitoring of heart rate, blood pressure, respiratory rate, and oxygen saturation during the Post-Anesthesia Care Unit stay. Adverse events will be recorded and graded according to Common Terminology Criteria for Adverse Events. A Data Safety Monitoring Committee will review safety data at regular intervals. Pre-specified stopping rules include rates of serious adverse events exceeding 5% in either group or significant imbalances in adverse events between groups.

Study Duration Patient enrollment is expected to occur over 18 to 24 months. Each patient will be followed for 24 hours after surgery. Total study duration is anticipated to be 30 months including enrollment, follow-up, data analysis, and manuscript preparation.

ELIGIBILITY:
Inclusion Criteria:

Age 6 months to 6 years

Scheduled bilateral myringotomy with tube placement

ASA physical status I-II

Parent/guardian consent

Exclusion Criteria:

* Allergy to study medications (fentanyl, ketorolac, bupivacaine)

Renal impairment or contraindication to ketorolac

Bleeding disorder or anticoagulation

Significant obstructive sleep apnea (AHI >10)

Concurrent surgical procedures beyond BMT

Unilateral procedure only

Recent analgesic use (<24 hours)

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Moderate-to-Severe Pain (FLACC Score ≥4) During PACU Stay | From PACU admission to PACU discharge, up to 1 hour
  Number of participants experiencing at least one FLACC (Face, Legs, Activity, Cry, Consolability) scale score of 4 or greater during Post-Anesthesia Care Unit stay. FLACC is a validated behavioral pain assessment tool scored 0-10, with scores ≥4 indicating moderate-to-severe pain. FLACC scores assessed every 15 minutes during PACU stay.

SECONDARY OUTCOMES:
Highest FLACC Pain Score During PACU Stay | From PACU admission to meeting PACU discharge criteria
Number of Participants Requiring Rescue Analgesia | From PACU admission to meeting PACU discharge criteria
  Number of participants requiring at least one dose of rescue analgesic medication for FLACC score ≥4
Number of Participants with Respiratory Depression | From PACU admission to meeting PACU discharge criteria
  Number of participants with oxygen saturation below 95% requiring intervention (supplemental oxygen, stimulation, or airway repositioning)
Number of Participants with Postoperative Nausea and Vomiting | From PACU admission to meeting PACU discharge criteria
  Number of participants experiencing at least one episode of nausea or vomiting
Number of Participants with Emergence Agitation | From PACU admission to meeting PACU discharge criteria
  Number of participants with Pediatric Anesthesia Emergence Delirium (PAED) scale score ≥10, indicating clinically significant emergence agitation
PACU Length of Stay | From PACU admission to meeting PACU discharge criteria
  Duration in minutes from PACU admission to meeting discharge criteria
Parent Satisfaction with Pain Management | At 24 hours postoperatively
  Parent-reported satisfaction with pain management assessed on 5-point Likert scale (1=very dissatisfied to 5=very satisfied)
Need for additional analgesics at home | At 24 hours postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Children and Woman's Hospital, Mobile, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cook-Sather SD, Castella G, Zhang B, Mensinger JL, Galvez J, Wetmore RF. Principal Factors Associated With Ketorolac-Refractory Pain Behavior After Pediatric Myringotomy and Pressure Equalization Tube Placement: A Retrospective Cohort Study. Anesth Analg. 2020 Mar;130(3):730-739. doi: 10.1213/ANE.0000000000004226. PMID 31082971
- [Background] Voronov P, Tobin MJ, Billings K, Cote CJ, Iyer A, Suresh S. Postoperative pain relief in infants undergoing myringotomy and tube placement: comparison of a novel regional anesthetic block to intranasal fentanyl--a pilot analysis. Paediatr Anaesth. 2008 Dec;18(12):1196-201. doi: 10.1111/j.1460-9592.2008.02789.x. PMID 19076574
- [Result] Cohen WG, Zhang B, Lee DR, Ampah SB, Sobol SE, Cook-Sather SD. Middle Ear Condition at the Time of Pediatric Myringotomy Tube Placement: Pain Associations Following Intraoperative Fentanyl/Ketorolac and Seasonal Variation. Anesth Analg. 2023 May 1;136(5):975-985. doi: 10.1213/ANE.0000000000006230. Epub 2022 Nov 2. PMID 36525380